CLINICAL TRIAL: NCT06790771
Title: Acute Effect of Supplement Containing L-Arginine on Appetite Suppression and GLP-1 Induction
Brief Title: Effect of Supplement on Appetite and GLP-1
Acronym: GLP-1 Suppleme
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Christian University (Other)
Collaborators: Healthrite Partners (Unknown); GMT Nutrition, LLC (Unknown)
Responsible Party: Principal Investigator, Elisa Marroquin, Assistant Professor, Texas Christian University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: TCU GLP-1 Study
Record Dates: First submitted 2025-01-07; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Hunger
Keywords: Hunger; GLP-1; Satiety; Supplement

STUDY DESIGN:
Intervention Model Description: Each participant will undergo the three experimental conditions in random order. Each intervention will be separated by a wash out period of 1 week.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a triple-blinded study, meaning neither the participants, researchers, nor analysts will know which condition is being tested during each visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): The placebo arm serves as the control condition, using a ~5 g powder with no active ingredients. Participants follow the same protocol as the other arms, including an 8-hour fasting period, baseline blood sample collection, and consumption of the placebo before a 60-minute rest. They then eat the standardized meal ad libitum (within a time window of 30 minutes), with blood samples collected at the eight time points and hunger levels assessed using the 7-point scale. The placebo arm is expected to show minimal or no effect on GLP-1 secretion and hunger suppression, providing a baseline for comparison against the two active supplement doses.
  Interventions: Dietary Supplement: Placebo
- High Dose Supplement (Experimental): In the high-dose supplement arm, participants consume approximately 10 grams of the nutritional supplement, which contains 9,000 mg of L-arginine, 200 mg of resveratrol, 500 mg of tart cherry, and 100 mg of vitamin C. After an 8-hour fasting period, participants visit the lab, where a baseline blood sample is collected before supplement consumption. They then rest for 60 minutes to allow absorption and subsequently eat a standardized meal (Bertolli Chicken Alfredo pasta bake) ad libitum within 30 minutes. Blood samples are collected at eight time points, and hunger levels are measured using a 7-point satiety scale. This arm is expected to show the most pronounced effects on GLP-1 secretion and hunger suppression compared to the other arms, highlighting the potential efficacy of a high-dose intervention.
  Interventions: Dietary Supplement: High Dose Supplement
- Low Dose Supplement (Experimental): In the low-dose supplement arm, participants consume approximately 5 grams of the supplement, consisting of 4,500 mg of L-arginine, 100 mg of resveratrol, 250 mg of tart cherry, and 50 mg of vitamin C. As in the high-dose arm, participants arrive after fasting for 8 hours, provide a baseline blood sample, and consume the supplement before a 60-minute rest. Following the rest period, they eat the same standardized meal ad libitum within a time window of 30 minutes. Blood samples are again taken at eight time points, and hunger levels are recorded using the same scale. This arm evaluates whether a reduced dose of the supplement provides moderate effects on GLP-1 secretion and hunger suppression, potentially identifying a lower effective dose.
  Interventions: Dietary Supplement: Low Dose Supplement

INTERVENTIONS:
Dietary Supplement: High Dose Supplement — Participants in this intervention receive approximately 10 grams of the supplement, containing 9,000 mg of L-arginine, 200 mg of resveratrol, 500 mg of tart cherry, and 100 mg of vitamin C. The supplement is consumed in powdered form after an 8-hour fasting period. Following a 60-minute rest, participants eat an ad libitum meal to assess the supplement's effect on hunger and food intake. Blood samples are collected at eight specific time points to measure metabolic markers, including GLP-1 levels, while hunger is tracked using a 7-point satiety scale. This intervention aims to determine the effects of a high dose of the supplement on appetite suppression and metabolic responses.
  Arms: High Dose Supplement
Dietary Supplement: Low Dose Supplement — In this intervention, participants consume approximately 5 grams of the supplement, which contains 4,500 mg of L-arginine, 100 mg of resveratrol, 250 mg of tart cherry, and 50 mg of vitamin C. The protocol mirrors that of the high-dose intervention: participants arrive after fasting for 8 hours, consume the supplement, rest for 60 minutes, and eat the standardized ad libitum meal. Blood samples are taken at the same eight time points to assess metabolic responses, and hunger levels are measured using the same satiety scale. This intervention investigates whether a lower dose of the supplement can still significantly affect hunger and GLP-1 secretion.
  Arms: Low Dose Supplement
Dietary Supplement: Placebo — The placebo intervention involves participants consuming a ~5 g inert powder with no active ingredients. Participants follow the same protocol as the other two interventions, including fasting, baseline blood collection, supplement (placebo) consumption, a 60-minute rest, and an ad libitum meal. Blood samples are collected at eight time points, and hunger levels are assessed with the 7-point scale. This intervention serves as a control, helping to determine whether observed effects in the other two interventions are attributable to the active supplement ingredients.
  Arms: Placebo

SUMMARY:
Study Summary

The goal of this study is to understand whether a dietary supplement containing L-arginine, resveratrol, tart cherry, and vitamin C reduces hunger and increases the release of GLP-1, a hormone associated with appetite suppression and improved glucose regulation. The study will also explore the metabolic effects of the supplement.

Main Questions:

1. Does the supplement reduce hunger more effectively than a placebo?
2. Does it enhance GLP-1 release in individuals with overweight or obesity?

Participants:

* Age: 18-60 years
* Body Mass Index (BMI): 25-40 kg/m²
* Total participants: 25
* Must maintain usual eating and activity habits during the study.

Study Design:

* Conditions Tested: High-dose supplement, low-dose supplement, and placebo.
* Participants will undergo three separate 2-hour lab visits, each after fasting for 8 hours.
* During each visit:
* Consume the assigned supplement or placebo.
* Eat a standardized meal after a 60-minute rest.
* Provide blood samples at eight time points to measure GLP-1 and other metabolic markers.
* Rate hunger using a 7-point scale.

Benefits and Risks:

* Benefits: Participants may not directly benefit, but the findings could lead to new appetite-suppressing supplements that aid in weight loss.
* Risks: Include discomfort from blood draws, possible gastrointestinal side effects from the supplement, and allergic reactions. Measures are in place to minimize these risks, such as pre-screening for allergies and using trained personnel for blood collection.

This study is triple-blinded, meaning neither the participants, researchers, nor analysts will know which condition is being tested during each visit. Data collected will be anonymized to protect participant privacy.

DETAILED DESCRIPTION:
Study Title:

Acute Effect of Supplement Containing L-Arginine on Appetite Suppression and GLP-1 Induction

Research Objectives:

The study aims to evaluate the effects of a dietary supplement containing L-arginine, resveratrol, tart cherry, and vitamin C on appetite suppression, GLP-1 hormone release, and associated metabolic outcomes in individuals with overweight or obesity.

Background:

GLP-1 (Glucagon-Like Peptide 1) plays a crucial role in regulating appetite and glucose homeostasis.

Condensed Background Information:

The combination of the following ingredients is hypothesized to have a synergistic effect, promoting satiety and improving metabolic health:

* L-arginine enhances GLP-1 secretion, improving glucose tolerance and reducing appetite.
* Resveratrol inhibits DPP-IV, extending the activity of GLP-1.
* Tart cherry supports metabolic regulation by enhancing nitric oxide availability and preventing arginine catabolism.
* Vitamin C acts as an antioxidant, supporting the efficacy of other components.

Participant Details:

* Number of Participants: 25
* Eligibility Criteria:
* Adults aged 18-60 years.
* BMI between 25 and 40 kg/m².
* Must maintain current diet and physical activity levels.

Exclusion Criteria:

* Significant weight change (>5%) in the last three months.
* Medical conditions like uncontrolled diabetes, kidney disease, thyroid disorders, or autoimmune diseases.
* Current use of medications or supplements affecting weight or GLP-1 levels.
* Pregnancy or lactation.

Study Design:

This is a randomized, triple-blinded, placebo-controlled study with three conditions:

* High-Dose Supplement (~10 g)
* Low-Dose Supplement (~5 g)
* Placebo (~5 g) Each participant will experience all three conditions in random order.

The timeline for the study involves:

* Pre-Session: 8-hour fasting before each visit.
* Arrival at the lab (Rickel Building, Rooms 256/259).
* Baseline blood sample collection.
* Administration of assigned supplement/placebo.
* 60-minute rest period.
* Consumption of a standardized meal (Bertolli Chicken Alfredo pasta bake) in isolation within a 30-minute window.
* Collection of additional blood samples at eight-time points
* Measurement of hunger using a 7-point scale.

Study Procedures

Blood Sampling:

* 7 mL samples collected at each time point for metabolic analysis (e.g., glucose, insulin, GLP-1).
* Total blood volume: 168 mL per participant across all sessions.
* Samples will be analyzed for metabolic markers in Dr. Ryan Porter's lab.

Satiety Measurement:

Participants will rate hunger levels at each blood draw using a scale from "Extremely Hungry" to "Extremely Full."

Meal Intake:

An ad libitum meal is provided to assess the impact of supplementation on food consumption.

Risks and Mitigation

* Blood Draw Risks: Bruising, pain, infection, or dizziness. Managed by using trained personnel and aseptic techniques.
* Supplement Risks: Gastrointestinal discomfort and allergic reactions. Addressed by pre-screening participants for allergies. Emergency supplies will be available.
* Data Privacy Risks:

All data will be anonymized and stored securely to prevent breaches.

Expected Outcomes

The study aims to determine:

* If the supplement reduces hunger compared to a placebo.
* If it enhances GLP-1 release post-meal.
* If it improves other metabolic parameters (e.g., glucose, lipid profiles).

Data Handling:

All data will be anonymized and securely stored. Samples may be retained for up to 24 months for further research.

Statistical Analysis:

Data analysis will use ANOVA and Tukey's post-hoc tests in SPSS, with significance set at p<0.05.

Study Impact:

This research could contribute to developing effective nutritional interventions to support appetite regulation and weight management, benefiting individuals with obesity and/or metabolic disorders.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following conditions to be eligible for the study:

* Age: 18-60 years old.
* BMI (Body Mass Index): Between 25 and 40 kg/m².
* Diet and Activity Stability: Willing to maintain current dietary and physical activity habits for the duration of the study.

Exclusion Criteria:

Participants will be excluded from the study if any of the following conditions apply:

* Recent Weight Change: Lost or gained more than 5% of body weight in the last 3 months.
* Pregnancy or Lactation: Pregnant or breastfeeding women.
* Medical Conditions:

  * Kidney disease (Chronic Kidney Disease or End-Stage Renal Disease).
  * Herpes simplex.
  * Uncontrolled diabetes (HbA1c >7%).
  * Thyroid disorders or taking thyroid medications.
  * Type 1 diabetes.
  * Cushing syndrome.
  * Cirrhosis or hepatitis.
  * Chronic obstructive pulmonary disease (COPD).
  * Dementias.
  * Active autoimmune diseases (e.g., lupus, rheumatoid arthritis).
  * Crohn's disease or ulcerative colitis.
  * Celiac disease.
  * Allergies or Sensitivities:
  * Known allergies to any components of the supplement or standardized meal.
  * Medications: Currently taking any of the following:
* Supplements or medications for weight loss.
* Antihypertensive, antidiabetic, or antihyperlipidemic medications.
* Erectile dysfunction medications.
* Blood thinners (e.g., aspirin, warfarin).
* Medications containing nitric oxide or nitroglycerin.
* Drugs affecting GLP-1 levels, such as GLP-1 receptor agonists, insulin, certain antidepressants, or corticosteroids.

  * Substance Use: Evidence of illegal drug use, including marijuana.
  * Participation in Other Studies: Enrollment in another clinical trial that could interfere with the study outcomes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Appetite | 2 hours per session, measured during three separate sessions over three weeks.
  This measure tracks participants' subjective hunger levels using a validated 7-point satiety scale (ranging from "Extremely Hungry" to "Extremely Full"). Ratings will be recorded at each of the eight time points corresponding to blood sample collection to assess the effect of the supplement on appetite suppression.
Food Intake | Single meal during each session, measured in three sessions over three weeks.
  This measure evaluates the amount of food consumed during the ad libitum standardized meal provided at each session. Participants will eat until they feel comfortably full, and the total food intake will be weighed to assess the impact of the interventions on caloric consumption.
Blood Glucose | 2 hours per session, measured during three separate sessions over three weeks.
  This measure tracks changes in blood glucose concentrations at the same eight time points (baseline, 15, 30, 45, 60, 90, 105, and 120 minutes) as GLP-1 sampling. It evaluates the impact of the supplement on glucose regulation following supplementation and meal intake.

SECONDARY OUTCOMES:
Insulin Levels | 2 hours per session, measured during three separate sessions over three weeks.
  This measure examines the acute changes in circulating insulin levels at the same eight time points to determine the supplement's effect on insulin secretion and glucose metabolism.
Lipid Profile Levels | 2 hours per session, measured during three separate sessions over three weeks.
  This measure assesses changes in lipid markers, such as triglycerides and cholesterol, at the same eight time points. It evaluates the supplement's potential effects on postprandial lipid metabolism.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Specific IPD That Can Be Shared
  Demographic Data:
  * Age
  * Sex
  Anthropometric Data:
  - BMI
  Outcome Measures:
  * GLP-1 levels
  * Hunger ratings
  * Food intake data (grams or kcal)
  * Blood glucose levels
  * Insulin levels
  * Lipid profile markers
  Adverse Events or Side Effects:
  * Reports of gastrointestinal distress or other reactions to the supplement
  * Any issues related to blood sampling
  Session Attendance and Compliance:
  * Adherence to fasting requirements
  * Completion of all study sessions
  Conditions for Sharing IPD De-Identification: Investigators will remove all personal identifiers (e.g., name, contact information, date of birth).
  Data Aggregation: Investigators will aggregate data if necessary to prevent re-identification of participants.
  Access Control: Share data only with authorized researchers who request it or for peer-reviewed publications.
  Informed Consent: Investigators will ensure participants are aware and have agreed to the potential sharing of de-identified data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after the publication of the primary results and for up to 24 months following the completion of the study.
Access Criteria: Access to the Individual Participant Data (IPD) and supporting information will be granted to:
  Qualified Researchers: Academic or clinical researchers affiliated with recognized institutions who request the data for scientific purposes and demonstrate a legitimate interest in advancing the study's objectives.
  Regulatory Bodies and Sponsors: Regulatory agencies (e.g., IRB and IBC) and study sponsors (sponsors) may access de-identified data for verification, compliance, or reporting purposes.
  Journal Reviewers: Summary data and de-identified results may be shared during manuscript submission and peer review.
  What Will Be Shared?
  * De-identified GLP-1 levels, hunger ratings, food intake, glucose levels, insulin levels, lipid profiles, and session compliance data.
  * Supporting Documentation: study protocol, statistical analysis plan, and metadata necessary for interpreting the datasets.
  * Summarized outcomes (e.g., means, SD) for each intervention arm may also be shared.

REFERENCES:
- [Background] Lucotti P, Setola E, Monti LD, Galluccio E, Costa S, Sandoli EP, Fermo I, Rabaiotti G, Gatti R, Piatti P. Beneficial effects of a long-term oral L-arginine treatment added to a hypocaloric diet and exercise training program in obese, insulin-resistant type 2 diabetic patients. Am J Physiol Endocrinol Metab. 2006 Nov;291(5):E906-12. doi: 10.1152/ajpendo.00002.2006. Epub 2006 Jun 13. PMID 16772327
- [Background] Dashtabi A, Mazloom Z, Fararouei M, Hejazi N. Oral L-Arginine Administration Improves Anthropometric and Biochemical Indices Associated With Cardiovascular Diseases in Obese Patients: A Randomized, Single Blind Placebo Controlled Clinical Trial. Res Cardiovasc Med. 2015 Dec 29;5(1):e29419. doi: 10.5812/cardiovascmed.29419. eCollection 2016 Feb. PMID 26889456
- [Background] Rogers DR, Lawlor DJ, Moeller JL. Vitamin C Supplementation and Athletic Performance: A Review. Curr Sports Med Rep. 2023 Jul 1;22(7):255-259. doi: 10.1249/JSR.0000000000001083. PMID 37417662
- [Background] Ceriello A, Novials A, Ortega E, Canivell S, Pujadas G, La Sala L, Bucciarelli L, Rondinelli M, Genovese S. Vitamin C further improves the protective effect of GLP-1 on the ischemia-reperfusion-like effect induced by hyperglycemia post-hypoglycemia in type 1 diabetes. Cardiovasc Diabetol. 2013 Jun 27;12:97. doi: 10.1186/1475-2840-12-97. PMID 23806096
- [Background] Hooper DR, Orange T, Gruber MT, Darakjian AA, Conway KL, Hausenblas HA. Broad Spectrum Polyphenol Supplementation from Tart Cherry Extract on Markers of Recovery from Intense Resistance Exercise. J Int Soc Sports Nutr. 2021 Jun 14;18(1):47. doi: 10.1186/s12970-021-00449-x. PMID 34126996
- [Background] Bordage S, Pham TN, Zedet A, Gugglielmetti AS, Nappey M, Demougeot C, Girard-Thernier C. Investigation of Mammal Arginase Inhibitory Properties of Natural Ubiquitous Polyphenols by Using an Optimized Colorimetric Microplate Assay. Planta Med. 2017 May;83(7):647-653. doi: 10.1055/s-0042-118711. Epub 2016 Oct 24. PMID 27776374
- [Background] Kim DW, Jung DH, Sung J, Min IS, Lee SJ. Tart Cherry Extract Containing Chlorogenic Acid, Quercetin, and Kaempferol Inhibits the Mitochondrial Apoptotic Cell Death Elicited by Airborne PM10 in Human Epidermal Keratinocytes. Antioxidants (Basel). 2021 Mar 13;10(3):443. doi: 10.3390/antiox10030443. PMID 33805724
- [Background] Huang PK, Lin SR, Chang CH, Tsai MJ, Lee DN, Weng CF. Natural phenolic compounds potentiate hypoglycemia via inhibition of Dipeptidyl peptidase IV. Sci Rep. 2019 Oct 30;9(1):15585. doi: 10.1038/s41598-019-52088-7. PMID 31666589
- [Background] Hurt RT, Ebbert JO, Schroeder DR, Croghan IT, Bauer BA, McClave SA, Miles JM, McClain CJ. L-arginine for the treatment of centrally obese subjects: a pilot study. J Diet Suppl. 2014 Mar;11(1):40-52. doi: 10.3109/19390211.2013.859216. Epub 2014 Jan 10. PMID 24409974
- [Background] Amin A, Neophytou C, Thein S, Martin NM, Alamshah A, Spreckley E, Bloom SR, Murphy KG. L-Arginine Increases Postprandial Circulating GLP-1 and PYY Levels in Humans. Obesity (Silver Spring). 2018 Nov;26(11):1721-1726. doi: 10.1002/oby.22323. PMID 30358156
- [Background] Clemmensen C, Smajilovic S, Smith EP, Woods SC, Brauner-Osborne H, Seeley RJ, D'Alessio DA, Ryan KK. Oral L-arginine stimulates GLP-1 secretion to improve glucose tolerance in male mice. Endocrinology. 2013 Nov;154(11):3978-83. doi: 10.1210/en.2013-1529. Epub 2013 Aug 19. PMID 23959939